CLINICAL TRIAL: NCT01787552
Title: A Phase Ib/II, Open-label, Multi-center, Dose-finding Study to Assess the Safety and Efficacy of the Oral Combination of LDE225 and INC424 (Ruxolitinib) in Patients With Myelofibrosis
Brief Title: A Phase Ib/II Dose-finding Study to Assess the Safety and Efficacy of LDE225 + INC424 in Patients With MF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDE225X2116; 2012-004023-20 (EudraCT Number)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Primary Myelofibrosis; Thrombocytosis; Essential Thrombocythemia; Polycythemia Vera; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases; Blood Coagulation Disorders; Blood Platelet Disorders; Hemorrhagic Disorders
Keywords: Dose escalation; Maximum Tolerated Dose; MTD; Safety Expansion; Safety; Efficacy; Myelofibrosis; Post-polycythemia vera myelofbrosis (Post PV-PMF); Post essential thrombocythemia myelofibrosis (Post ET-MF); Primary myelofibrosis (PMF); Intermediate risk myelofibrosis; High risk myelofibrosis; Combination Treatment; Hedgehog Signaling Pathway; Smoothened inhibitor; JAK inhibitor
MeSH Terms: conditions — Primary Myelofibrosis; Thrombocytosis; Thrombocythemia, Essential; Polycythemia Vera; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases; Blood Coagulation Disorders; Blood Platelet Disorders; Hemorrhagic Disorders | interventions — sonidegib; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDE225 + INC424 (Experimental): LDE225 and INC424 in combination
  Interventions: Drug: LDE225; Drug: INC424

INTERVENTIONS:
Drug: LDE225
Drug: INC424

SUMMARY:
The purpose of this phase Ib/II clinical trial was to: a) evaluate the safety of the co-administration of LDE225 and INC424 in myelofibrosis patients and establish a maximum tolerated dose and/or Recommended Phase II dose of the combination and b) to assess the efficacy of the co-administration of LDE225 and INC424 on spleen volume reduction.

DETAILED DESCRIPTION:
The study is considered to have been completed because the participants completed the study as per study design at the time of trial termination. If participants were already in extension phase until discontinuation criteria were met or alternative setting was available, they were considered as completed. The study was terminated due to one of the compounds being divested.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PMF per 2008 WHO criteria, post-PV MF or post-ET MF per IWG-MRT criteria.
* Ineligible or unwilling to undergo stem cell transplantion.
* PLT counts > or = 75X 10^9/L not reached with the aid of transfusions.
* ECOG performance status ≤ 2.
* Palpable splenomegaly defined as ≥ 5 cm below the left costal margin.
* Intermediate risk level 1 (1 prognostic factor which is not age), Intermediate risk level 2, or high risk.
* Active symptoms of MF as demonstrated by one symptom score of at least 5 (0 to10 point scale) or two symptom scores of at least 3 (0 to 10 point scale) on the MF Symptom Assessment Form (MFSAF).

Exclusion Criteria:

* Previous therapy with JAK or Smoothened inhibitors.
* Patient is currently on medications that interfere with coagulation (including warfarin) or platelet function with the exception of low dose aspirin (up to 100 mg) and LMWH.
* Impairment of GI function or GI disease that may significantly alter the absorption of INC424 or LDE225 (e.g., uncontrolled nausea, vomiting, diarrhea; malabsorption syndrome; small bowel resection).
* Splenic irradiation within 12 months prior to Screening.
* Pregnant or nursing women.
* WOCBP not using highly effective methods of contraception
* Sexually active males who refuse condom use
* Patients who have neuromuscular disorders (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis and spinal muscular atrophy) or are on concomitant treatment with drugs that are recognized to cause rhabdomyolysis, such as HMG CoA inhibitors (statins), clofibrate and gemfibrozil. Pravastatin may be used if necessary, with extra caution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05-08 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- Australia (2):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
- Novartis Investigative Site, Leuven, Belgium
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Roskilde, Denmark
- Novartis Investigative Site, Marseille, France
- Germany (2):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Magdeburg
- Novartis Investigative Site, Galway, Ireland
- Italy (2):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Reggio Calabria, RC
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Rotterdam
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- United Kingdom (2):
  - Novartis Investigative Site, Glasgow, Scotland
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Gupta V, Wolleschak D, Hasselbalch H, Vannucchi AM, Koschmieder S, Cervantes F, Li Y, Dong T, Wroclawska M, Bharathy S, Harrison C. Safety and efficacy of the combination of sonidegib and ruxolitinib in myelofibrosis: a phase 1b/2 dose-finding study. Blood Adv. 2020 Jul 14;4(13):3063-3071. doi: 10.1182/bloodadvances.2019001212. PMID 32634234

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 50 subjects were enrolled in the study, of which 23 subjects were enrolled in Phase Ib part of dose-escalation phase and 27 subjects were enrolled in Phase Ib dose-expansion phase and Phase II Stage 1.
Pre-assignment Details: A total of 50 subjects were enrolled in the study, of which 23 subjects were enrolled in Phase Ib part of dose-escalation phase and 27 subjects were enrolled in Phase Ib dose-expansion phase and Phase II Stage 1.
Groups:
- LDE225 400mg + INC424 10 mg (Dose Escalation Phase): Participants who took a combination of LDE225 400mg and INC424 10mg in the dose escalation phase.
- LDE225 400mg + INC424 15 mg (Dose Escalation Phase): Participants who took a combination of LDED225 400mg and INC424 15mg in the dose escalation phase
- LDE225 400mg + INC424 20mg (Dose Escalation Phase): Participants who took a combination of LDE225 400mg and INC424 20mg in the dose escalation phase.
- LDED225 400mg + INC424 20mg (Dose Expansion Phase): Participants who took a combination of LDED225 400mg and INC424 20mg in the dose expansion phase
Period: Overall Study
Arm/Group | LDE225 400mg + INC424 10 mg (Dose Escalation Phase) | LDE225 400mg + INC424 15 mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Started | 8 | 10 | 5 | 27
Completed | 0 | 1 | 0 | 0
Not Completed | 8 | 9 | 5 | 27
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 4
Not completed — Physician Decision | 2 | 2 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Adverse Event | 2 | 5 | 2 | 16
Not completed — Study terminated by Sponsor | 0 | 0 | 1 | 3
Not completed — Progressive Disease | 2 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LDE225 400mg + INC424 10 mg (Dose Escalation Phase) | LDE225 400mg + INC424 15 mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase) | Total
Number analyzed (Participants) | 8 | 10 | 5 | 27 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.9 (5.19) | 59.9 (11.59) | 64.6 (13.18) | 67.4 (10.02) | 66.2 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 1 | 8 | 15
  Male | 7 | 5 | 4 | 19 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 10 | 5 | 26 | 47
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) (Phase 1b)
Description: A dose-limiting toxicity (DLT) was defined as an adverse event or abnormal laboratory value assessed as unrelated to disease progression, inter-current illness, or concomitant medications that met certain criteria as defined in the protocol.
Time Frame: 6 weeks (42 days)
Population: Safety Analysis Set (SAS) included all participants in Phase Ib & Phase II who received at least 1 dose of LDE225 and/or INC424 & had at least 1 valid post-baseline safety assessment. DLT was measured in the Phase Ib dose escalation & expansion phase, as part of the primary outcome. All participants in the safety set were considered for toxicities.
Measure: Count of Participants; unit: Participants
Groups:
- LDE225 400mg + INC424 10mg (Dose Escalation Phase): Participants who took a combination of LDE225 400mg and INC424 10mg in the dose escalation phase.
- LDE225 400mg + INC424 15mg (Dose Escalation Phase): Participants who took a combination of LDED225 400mg and INC424 15mg in the dose escalation phase
- LDE225 400mg + INC424 20mg (Dose Escalation Phase): Participants who took a combination of LDED225 400mg and INC424 20mg in the dose escalation phase
Arm/Group | LDE225 400mg + INC424 10mg (Dose Escalation Phase) | LDE225 400mg + INC424 15mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 8 | 10 | 5 | 27
Participants
  Blood creatine phosphokinase increased | 0 | 2 | 0 | 1

2. Primary Outcome: Percentage of Patients Achieving >= 35% Reduction in Spleen Volume in Phase Ib Expansion and Phase II Stage 1
Description: Reduction in spleen volume as measured by magnetic resonance imaging/Cat Scan (MRI/CT) in Phase Ib expansion and Phase II Stage 1 patients
Time Frame: Week 24 and Week 48
Population: The Full Analysis Set (FAS) comprised all subjects in Phase Ib and Phase II who received at least one dose of LDE225 and/or INC424. The data disclosed includes only participants from Phase Ib dose expansion phase and Ph II Stage 1. This data does not include dose escalation Phase Ib participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 27
Percentage of Participants
  Week 24 | 44.4
  Week 48 | 29.6

3. Secondary Outcome: Phase Ib and Phase II: LDE225: Plasma Pharmacokinetics (PK) Parameter: Area Under the Curve(AUC0-24h)
Description: Plasma Concentration Time Curve: AUC0-24h: Area under the concentration-time curve from time zero to 24 hours extrapolate from AUClast[mass x time x volume-1]
Time Frame: 0, 0.5, 1. 1.5, 2, 4, 6, 8 hrs on Week 1 Day 1 & Week 9 Day 1
Population: The Pharmacokinetic Analysis set (PAS) consisted of all subjects in Phase Ib and Phase II who received at least one (full or partial) dose of LDE225 and/or INC424 and provided at least one evaluable PK blood sample for LDE225 and/or INC424.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | LDE225 400mg + INC424 10mg (Dose Escalation Phase) | LDE225 400mg + INC424 15mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 8 | 10 | 5 | 27
ng*hr/mL
  LDE225 (Week 1, Day 1) (n=6,10,4,24): number analyzed (Participants) | 6 | 10 | 4 | 24
  LDE225 (Week 1, Day 1) (n=6,10,4,24) | 2680 (33.1) | 1900 (100.4) | 1090 (84.0) | 2060 (78.7)
  LDE225 (Week 9, Day 1) (n=6,6,4,14): number analyzed (Participants) | 6 | 6 | 4 | 14
  LDE225 (Week 9, Day 1) (n=6,6,4,14) | 15500 (31.8) | 13000 (66.8) | 17100 (30.8) | 14500 (45.4)

4. Secondary Outcome: Phase Ib and Phase II: INC424: PK Parameters: Area Under the Curve for AUC0-12h, AUCinf & AUClast
Description: AUC0-12h: Area under the concentration-time curve from time zero to 12 hours extrapolate from AUClast[mass x time x volume-1]. AUCinf: Area under the concentration-time curve from time zero to infinity with extrapolation of the terminal phase [mass x time x volume-1]. AUClast: Area under the concentration-time curve from time zero to the time of last measurable concentration [mass x time x volume-1].
Time Frame: 0, 0.5, 1. 1.5, 2, 4, 6, 8 hrs on Week 1 Day 1 & Week 9 Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | LDE225 400mg + INC424 10mg (Dose Escalation Phase) | LDE225 400mg + INC424 15mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 8 | 10 | 5 | 27
ng*hr/mL
  AUC0-12h: Wk1 Day 1 (n=8,10,5,25): number analyzed (Participants) | 8 | 10 | 5 | 25
  AUC0-12h: Wk1 Day 1 (n=8,10,5,25) | 473 (29.5) | 805 (45.6) | 1130 (23.0) | 1190 (41.0)
  AUC0-12h: Wk 9 Day 1 (n=8,9,4,20): number analyzed (Participants) | 8 | 9 | 4 | 20
  AUC0-12h: Wk 9 Day 1 (n=8,9,4,20) | 489 (42.5) | 835 (46.6) | 962 (23.7) | 1230 (42.4)
  AUCinf: Wk1 Day 1 (n=7,9,4,16): number analyzed (Participants) | 7 | 9 | 4 | 16
  AUCinf: Wk1 Day 1 (n=7,9,4,16) | 466 (30.9) | 789 (46.1) | 1140 (28.0) | 1130 (47.7)
  AUCinf: Wk 9 Day 1 (n=8,9,3,15): number analyzed (Participants) | 8 | 9 | 3 | 15
  AUCinf: Wk 9 Day 1 (n=8,9,3,15) | 498 (43.1) | 867 (48.7) | 978 (29.5) | 1140 (43.0)
  AUClast: Wk1 Day 1 (n=8,10,5,26): number analyzed (Participants) | 8 | 10 | 5 | 26
  AUClast: Wk1 Day 1 (n=8,10,5,26) | 443 (26.2) | 730 (39.7) | 1030 (20.8) | 1070 (38.6)
  AUClast: Wk 9 Day 1 (n=8,9,4,20): number analyzed (Participants) | 8 | 9 | 4 | 20
  AUClast: Wk 9 Day 1 (n=8,9,4,20) | 460 (44.3) | 776 (43.9) | 891 (24.3) | 1130 (38.6)

5. Secondary Outcome: Phase Ib and Phase II: LDE225 & INC424: PK Parameter: Maximum Plasma Concentration (Cmax)
Description: Cmax: Maximum observed plasma concentration after drug administration [mass x volume-
  1].
Time Frame: 0, 0.5, 1. 1.5, 2, 4, 6, 8 hrs on Week 1 Day 1 & Week 9 Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | LDE225 400mg + INC424 10mg (Dose Escalation Phase) | LDE225 400mg + INC424 15mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 8 | 10 | 5 | 27
ng/mL
  LDE225 (Week 1, Day 1) (n=6,10,5,26): number analyzed (Participants) | 6 | 10 | 5 | 26
  LDE225 (Week 1, Day 1) (n=6,10,5,26) | 311 (35.1) | 221 (103.4) | 161 (94.9) | 251 (83.4)
  LDE225 (Week 9, Day 1) (n=8,8,5,20): number analyzed (Participants) | 8 | 8 | 5 | 20
  LDE225 (Week 9, Day 1) (n=8,8,5,20) | 879 (38.0) | 720 (57.5) | 959 (39.4) | 951 (51.1)
  INC424 (Week 1, Day 1) (n=8,10,5,27) | 154 (29.0) | 244 (40.4) | 351 (27.7) | 338 (40.1)
  INC424 (Week 9, Day 1) (n=8,9,4,20): number analyzed (Participants) | 8 | 9 | 4 | 20
  INC424 (Week 9, Day 1) (n=8,9,4,20) | 168 (38.8) | 269 (33.2) | 281 (36.5) | 350 (36.0)

6. Secondary Outcome: Phase Ib and Phase II: LDE225 & INC424: Plasma PK Parameter: Time to Maximum Plasma Concentration (Tmax)
Description: Tmax: Time to reach Cmax [time]
Time Frame: 0, 0.5, 1. 1.5, 2, 4, 6, 8 hrs on Week 1 Day 1 & Week 9 Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | LDE225 400mg + INC424 10mg (Dose Escalation Phase) | LDE225 400mg + INC424 15mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 8 | 10 | 5 | 27
hour (hr)
  LDE225 (Week 1, Day 1) (n=6,10,5,26): number analyzed (Participants) | 6 | 10 | 5 | 26
  LDE225 (Week 1, Day 1) (n=6,10,5,26) | 3.01 [2.00 to 4.00] | 2.08 [1.50 to 4.22] | 2.00 [1.50 to 8.00] | 2.00 [1.00 to 6.00]
  LDE225 (Week 9, Day 1) (n=8,8,5,20): number analyzed (Participants) | 8 | 8 | 5 | 20
  LDE225 (Week 9, Day 1) (n=8,8,5,20) | 1.79 [0.170 to 4.00] | 2.00 [1.50 to 4.00] | 2.00 [1.50 to 6.00] | 3.21 [1.50 to 23.9]
  INC424 (Week 1, Day 1) (n=8,10,5,27) | 0.500 [0.500 to 2.00] | 0.575 [0.330 to 2.03] | 0.500 [0.500 to 0.970] | 0.580 [0.420 to 4.00]
  INC424 (Week 9, Day 1) (n=8,9,4,20): number analyzed (Participants) | 8 | 9 | 4 | 20
  INC424 (Week 9, Day 1) (n=8,9,4,20) | 0.875 [0.170 to 1.50] | 0.500 [0.500 to 1.52] | 1.00 [0.500 to 1.00] | 1.00 [0.330 to 2.00]

7. Secondary Outcome: Phase Ib and Phase II: LDE225 & INC424:: Plasma Pharmacokinetics (PK) Parameters: Area Under the Curve(CL/F)
Description: CL/F: Apparent total plasma clearance of drug after oral administration [volume x time-1]
Time Frame: 0, 0.5, 1. 1.5, 2, 4, 6, 8 hrs on Week 1 Day 1 & Week 9 Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: L/hr
Arm/Group | LDE225 400mg + INC424 10mg (Dose Escalation Phase) | LDE225 400mg + INC424 15mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 8 | 10 | 5 | 27
L/hr
  LDE225 (Week 1, Day 1) (n=5,5,1,12): number analyzed (Participants) | 5 | 5 | 1 | 12
  LDE225 (Week 1, Day 1) (n=5,5,1,12) | 145 [120 to 166] | 238 [53.7 to 508] | 727 [727 to 727] | 122 [46.2 to 525]
  LDE225 (Week 9, Day 1) (n=6,6,4,14): number analyzed (Participants) | 6 | 6 | 4 | 14
  LDE225 (Week 9, Day 1) (n=6,6,4,14) | 27.8 [14.9 to 35.7] | 34.5 [12.9 to 62.3] | 25.1 [15.4 to 30.9] | 27.0 [12.6 to 56.9]
  INC424 (Week 1, Day 1) (n=7,9,4,16): number analyzed (Participants) | 7 | 9 | 4 | 16
  INC424 (Week 1, Day 1) (n=7,9,4,16) | 23.8 [12.2 to 26.9] | 18.7 [9.04 to 39.0] | 16.5 [13.3 to 25.6] | 16.9 [7.54 to 35.0]
  INC424 (Week 9, Day 1) (n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Phase Ib and Phase II: Percentage of Participants With Fibrosis Grade Assessed by Bone Marrow Histomorphology, by Time and Treatment in Phase Ib and Phase II Stage 1
Description: The number of patients experiencing improvement in their bone marrow fibrosis by at least one grade and assessment of cellularity.
Time Frame: Baseline, Week 25 Day 1 (Week 24), Week 49 Day 1 (Week 48)
Population: The Full Analysis Set (FAS) comprised all subjects in Phase Ib and Phase II who received at least one dose of LDE225 and/or INC424.
Measure: Number; unit: Percentage of Participants
Arm/Group | LDE225 400mg + INC424 10mg (Dose Escalation Phase) | LDE225 400mg + INC424 15mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 8 | 10 | 5 | 27
Percentage of Participants
  Baseline, grade 0 (n=0,0,0,1): number analyzed (Participants) | 0 | 0 | 0 | 1
  Baseline, grade 0 (n=0,0,0,1) |  |  |  | 3.7
  Baseline, grade 1 (n=0,1,0,4): number analyzed (Participants) | 0 | 1 | 0 | 4
  Baseline, grade 1 (n=0,1,0,4) |  | 10.0 |  | 14.8
  Baseline, grade 2 (n=4,6,3,8): number analyzed (Participants) | 4 | 6 | 3 | 8
  Baseline, grade 2 (n=4,6,3,8) | 50.0 | 50.0 | 60.0 | 29.6
  Baseline, grade 3 (n=3,3,0,8): number analyzed (Participants) | 3 | 3 | 0 | 8
  Baseline, grade 3 (n=3,3,0,8) | 37.5 | 30.0 |  | 29.6
  Baseline, missing grade (n=1,0,2,6): number analyzed (Participants) | 1 | 0 | 2 | 6
  Baseline, missing grade (n=1,0,2,6) | 12.5 |  | 40.0 | 22.2
  Week 25 Day 1, grade 1 (n=1,1,0,1): number analyzed (Participants) | 1 | 1 | 0 | 1
  Week 25 Day 1, grade 1 (n=1,1,0,1) | 12.5 | 10.0 |  | 3.7
  Week 25 Day 1, grade 2 (n=0,3,2,7): number analyzed (Participants) | 0 | 3 | 2 | 7
  Week 25 Day 1, grade 2 (n=0,3,2,7) |  | 30.0 | 40.0 | 25.9
  Week 25 Day 1, grade 3 (n=5,4,1,5): number analyzed (Participants) | 5 | 4 | 1 | 5
  Week 25 Day 1, grade 3 (n=5,4,1,5) | 62.5 | 40.0 | 20.0 | 18.5
  Week 25 Day 1, missing grade (n=2,2,2,14): number analyzed (Participants) | 2 | 2 | 2 | 14
  Week 25 Day 1, missing grade (n=2,2,2,14) | 25.0 | 20.0 | 40.0 | 51.9
  Week 49 Day 1, grade 0 (n=0,0,0,1): number analyzed (Participants) | 0 | 0 | 0 | 1
  Week 49 Day 1, grade 0 (n=0,0,0,1) |  |  |  | 3.7
  Week 49, Day 1 grade 1 (n=0,0,0,1): number analyzed (Participants) | 0 | 0 | 0 | 1
  Week 49, Day 1 grade 1 (n=0,0,0,1) |  |  |  | 3.7
  Week 49 Day 1, grade 2 (n=0,1,1,2): number analyzed (Participants) | 0 | 1 | 1 | 2
  Week 49 Day 1, grade 2 (n=0,1,1,2) |  | 10.0 | 20.0 | 7.4
  Week 49 Day 1, grade 3 (n=2,2,2,3): number analyzed (Participants) | 2 | 2 | 2 | 3
  Week 49 Day 1, grade 3 (n=2,2,2,3) | 25.0 | 20.0 | 40.0 | 11.1
  Week 49 Day 1, missing grade (n=6,7,2,20): number analyzed (Participants) | 6 | 7 | 2 | 20
  Week 49 Day 1, missing grade (n=6,7,2,20) | 75.0 | 70.0 | 40.0 | 74.1

9. Secondary Outcome: Phase Ib and Phase ll: Summary of JAK2V617F Allele Burden by Visit and Treatment in Phase Ib and Phase II Stage 1
Description: Phase Ib and Phase ll: Change in Pharmacodynamic Biomarkers: JAK2V617F allele burden
Time Frame: Baseline, Week 25 Day 1 (Week 24), Week 49 Day 1 (Week 48)
Population: The Biomarker Analysis Set (BAS) consisted of all subjects in Phase Ib and Phase II who received at least one (full or partial) dose of LDE225 and/or INC424 and provided at least one evaluable biomarker sample.
Measure: Median (Full Range); unit: Percentage of JAK allele burden mutation
Arm/Group | LDE225 400mg + INC424 10mg (Dose Escalation Phase) | LDE225 400mg + INC424 15mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 8 | 10 | 5 | 27
Percentage of JAK allele burden mutation
  Baseline | 84.7 [48.4 to 95.1] | 61.7 [2.5 to 92.1] | 88.3 [52.7 to 94.4] | 55.4 [2.5 to 93.5]
  Week 25 Day 1 (n=7,6,5,21): number analyzed (Participants) | 7 | 6 | 5 | 21
  Week 25 Day 1 (n=7,6,5,21) | 88.6 [49.8 to 94.1] | 48.0 [2.5 to 78.4] | 74.9 [52.1 to 89.6] | 43.8 [2.5 to 93.9]
  Week 49 Day 1 (n=4,3,4,13): number analyzed (Participants) | 4 | 3 | 4 | 13
  Week 49 Day 1 (n=4,3,4,13) | 86.0 [20.1 to 94.1] | 54.3 [2.5 to 80.0] | 75.7 [56.9 to 90.0] | 46.1 [2.5 to 85.6]

10. Secondary Outcome: Phase Ib and Phase ll: Summary of Cytokine Levels in Pharmacodynamic for All Collected Biomarkers
Description: Summary of cytokine levels in Pharmacodynamic Biomarkers for all 26 collected at Week 25 Day 1 and Week 49 Day 1
Time Frame: Baseline, Week 25 Day 1 (Week 24), Week 49 Day 1 (Week 48)
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Arm/Group | LDE225 400mg + INC424 10mg (Dose Escalation Phase) | LDE225 400mg + INC424 15mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 8 | 10 | 5 | 27
ng/mL
  AFP: Week 25 Day 1 (Wk 25 D1) (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  AFP: Week 25 Day 1 (Wk 25 D1) (n=7,8,5,22) | 0.75 [0.3 to 2.5] | 0.79 [0.3 to 1.4] | 1.10 [0.3 to 2.2] | 0.49 [0.49 to 2.0]
  AFP: Week 49 Day 1 (WK25 D1) (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  AFP: Week 49 Day 1 (WK25 D1) (n=4,3,4,14) | 0.68 [0.3 to 1.6] | 0.60 [0.5 to 0.9] | 0.49 [0.49 to 1.1] | 0.49 [0.49 to 2.6]
  APOA-1: Week 25 Day 1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  APOA-1: Week 25 Day 1 (n=7,8,5,22) | 1.10 [0.7 to 1.7] | 1.65 [1.0 to 2.2] | 1.60 [1.2 to 1.6] | 2.10 [1.5 to 3.8]
  APOA-1: Week 49 Day 1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  APOA-1: Week 49 Day 1 (n=4,3,4,14) | 1.30 [0.9 to 1.5] | 1.50 [1.0 to 2.9] | 1.80 [1.6 to 2.6] | 2.05 [1.4 to 3.1]
  B2M: Week 25 Day 1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  B2M: Week 25 Day 1 (n=7,8,5,22) | 5.00 [2.8 to 7.4] | 3.15 [2.1 to 5.9] | 3.70 [2.4 to 5.2] | 3.15 [1.8 to 7.2]
  B2M: Week 49 Day 1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  B2M: Week 49 Day 1 (n=4,3,4,14) | 5.75 [4.5 to 11.0] | 4.60 [1.9 to 6.1] | 3.25 [2.4 to 4.4] | 3.00 [1.0 to 6.3]
  BDNF: Week 25 Day 1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  BDNF: Week 25 Day 1 (n=7,8,5,22) | 0.46 [0.0 to 2.0] | 0.85 [0.2 to 2.5] | 0.15 [0.1 to 0.4] | 0.55 [0.0 to 2.7]
  BDNF: Week 49 Day 1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  BDNF: Week 49 Day 1 (n=4,3,4,14) | 1.16 [0.3 to 2.4] | 0.19 [0.0 to 3.8] | 0.41 [0.0 to 5.6] | 0.52 [0.0 to 12.0]
  C Reactive Protein: Week 25 Day 1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  C Reactive Protein: Week 25 Day 1 (n=7,8,5,22) | 2.60 [1.0 to 16.0] | 2.70 [0.3 to 51.0] | 1.30 [0.1 to 4.1] | 4.50 [0.1 to 182.0]
  C Reactive Protein: Week 49 Day 1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  C Reactive Protein: Week 49 Day 1 (n=4,3,4,14) | 4.65 [0.4 to 9.0] | 2.40 [0.0 to 6.3] | 1.30 [0.7 to 2.5] | 0.79 [0.1 to 30.0]
  Carcinoembryyonic Antigen: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  Carcinoembryyonic Antigen: Wk 25 D1 (n=7,8,5,22) | 1.40 [0.3 to 58.0] | 1.20 [0.8 to 5.6] | 1.20 [0.3 to 3.4] | 1.80 [0.2 to 12.0]
  Carcinoembryyonic Antigen: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  Carcinoembryyonic Antigen: Wk 49 D1 (n=4,3,4,14) | 1.72 [0.8 to 3.7] | 1.20 [1.1 to 1.3] | 1.45 [0.5 to 2.6] | 1.80 [0.5 to 12.0]
  Cluster of. Diff 40: Wk 25 D1 (n=7,7,5,0): number analyzed (Participants) | 7 | 7 | 5 | 0
  Cluster of. Diff 40: Wk 25 D1 (n=7,7,5,0) | 1.90 [0.8 to 3.4] | 1.10 [0.6 to 1.6] | 0.91 [0.6 to 1.4] |
  Cluster of. Diff 40: Wk 49 D1 (n=4,2,0,0): number analyzed (Participants) | 4 | 2 | 0 | 0
  Cluster of. Diff 40: Wk 49 D1 (n=4,2,0,0) | 1.65 [0.9 to 2.4] | 1.3 [1.2 to 1.4] |  |
  Eotaxin1: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  Eotaxin1: Wk 25 D1 (n=7,8,5,22) | 155.00 [42.5 to 214.0] | 119.00 [42.5 to 429.0] | 101.00 [42.5 to 152.0] | 118.00 [58.5 to 294.0]
  Eotaxin1: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  Eotaxin1: Wk 49 D1 (n=4,3,4,14) | 136.00 [42.5 to 290.0] | 145.00 [58.5 to 622.0] | 157.00 [58.5 to 380.0] | 175.00 [58.5 to 360.0]
  ICAM1: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  ICAM1: Wk 25 D1 (n=7,8,5,22) | 266.00 [139.0 to 451.0] | 203.00 [137.0 to 339.0] | 168.00 [82.0 to 316.0] | 185.50 [93.0 to 324.0]
  ICAM1: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  ICAM1: Wk 49 D1 (n=4,3,4,14) | 321.00 [95.0 to 470.0] | 173.00 [94.0 to 193.0] | 152.50 [91.0 to 553.0] | 163.00 [92.0 to 310.0]
  IL10: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  IL10: Wk 25 D1 (n=7,8,5,22) | 9.30 [6.9 to 21.0] | 7.50 [3.4 to 11.0] | 3.40 [3.4 to 12.0] | 6.23 [4.1 to 29.0]
  IL10: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  IL10: Wk 49 D1 (n=4,3,4,14) | 8.10 [3.4 to 12.0] | 4.05 [3.4 to 18.0] | 11.00 [8.4 to 24.0] | 8.40 [4.1 to 28.0]
  IL18: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  IL18: Wk 25 D1 (n=7,8,5,22) | 292.00 [132.0 to 520.0] | 220.50 [108.0 to 907.0] | 445.00 [161.0 to 687.0] | 415.50 [127.0 to 1160.0]
  IL18: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  IL18: Wk 49 D1 (n=4,3,4,14) | 278.00 [146.0 to 606.0] | 199.00 [168.0 to 575.0] | 550.50 [313.0 to 1260.0] | 318.50 [134.0 to 886.0]
  IL1B: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  IL1B: Wk 25 D1 (n=7,8,5,22) | 3.30 [3.3 to 3.3] | 3.30 [3.3 to 4.3] | 3.30 [3.3 to 6.9] | 4.3 [4.3 to 16.0]
  IL1B: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  IL1B: Wk 49 D1 (n=4,3,4,14) | 3.30 [3.3 to 3.3] | 3.30 [3.3 to 4.3] | 4.3 [4.3 to 8.9] | 4.3 [4.3 to 10.0]
  IL1RN: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  IL1RN: Wk 25 D1 (n=7,8,5,22) | 130.00 [92.0 to 218.0] | 147.00 [85.0 to 496.0] | 114.00 [89.0 to 183.0] | 88.00 [63.0 to 328.0]
  IL1RN: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  IL1RN: Wk 49 D1 (n=4,3,4,14) | 98.00 [71.0 to 124.0] | 281.00 [29.5 to 782.0] | 88.00 [73.0 to 214.0] | 85.50 [29.5 to 162.0]
  IL6: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  IL6: Wk 25 D1 (n=7,8,5,22) | 4.70 [2.3 to 6.8] | 2.3 [2.3 to 6.3] | 2.3 [2.3 to 6.0] | 3.40 [3.4 to 11.0]
  IL6: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  IL6: Wk 49 D1 (n=4,3,4,14) | 3.48 [2.3 to 6.8] | 3.40 [2.3 to 4.7] | 3.40 [3.4 to 11.0] | 3.40 [3.4 to 7.3]
  IL8: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  IL8: Wk 25 D1 (n=7,8,5,22) | 28.00 [15.0 to 84.0] | 9.50 [7.2 to 74.0] | 15.00 [10.0 to 34.0] | 29.50 [6.9 to 280.0]
  IL8: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  IL8: Wk 49 D1 (n=4,3,4,14) | 18.50 [9.6 to 161.0] | 11.00 [8.4 to 19.0] | 58.50 [19.0 to 166.0] | 32.00 [3.1 to 261.0]
  Insulin: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  Insulin: Wk 25 D1 (n=7,8,5,22) | 2.70 [0.8 to 5.4] | 1.35 [0.6 to 3.3] | 2.30 [1.8 to 3.8] | 0.6 [0.6 to 8.9]
  Insulin: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  Insulin: Wk 49 D1 (n=4,3,4,14) | 2.90 [1.4 to 3.1] | 2.90 [0.6 to 4.9] | 1.65 [0.6 to 3.0] | 1.60 [0.6 to 14.0]
  LEP: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  LEP: Wk 25 D1 (n=7,8,5,22) | 1.50 [0.7 to 34.0] | 4.75 [1.2 to 30.0] | 6.00 [3.4 to 6.1] | 6.40 [1.2 to 49.0]
  LEP: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  LEP: Wk 49 D1 (n=4,3,4,14) | 3.45 [0.7 to 16.0] | 17.00 [2.7 to 29.0] | 5.95 [1.0 to 10.0] | 5.60 [3.3 to 28.0]
  Macro. Inflam. Prot-1 Beta: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  Macro. Inflam. Prot-1 Beta: Wk 25 D1 (n=7,8,5,22) | 491.00 [269.0 to 1160.0] | 375.50 [203.0 to 1260.0] | 410.00 [330.0 to 873.0] | 513.00 [190.0 to 1010.0]
  Macro. Inflam. Prot-1 Beta: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  Macro. Inflam. Prot-1 Beta: Wk 49 D1 (n=4,3,4,14) | 406.50 [242.0 to 758.0] | 487.00 [357.0 to 594.0] | 970.50 [489.0 to 1850.0] | 521.00 [159.0 to 1100.0]
  Macro.-derived Chemokine: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  Macro.-derived Chemokine: Wk 25 D1 (n=7,8,5,22) | 253.00 [43.0 to 599.0] | 274.00 [93.0 to 1040.0] | 516.00 [193.0 to 1100.0] | 254.00 [55.0 to 760.0]
  Macro.-derived Chemokine: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  Macro.-derived Chemokine: Wk 49 D1 (n=4,3,4,14) | 190.50 [9.5 to 852.0] | 327.00 [218.0 to 963.0] | 430.50 [132.0 to 801.0] | 212.00 [97.0 to 696.0]
  MPO: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  MPO: Wk 25 D1 (n=7,8,5,22) | 327.00 [127.0 to 1600.0] | 323.00 [134.0 to 3120.0] | 335.00 [134.0 to 3350.0] | 164.50 [63.0 to 1310.0]
  MPO: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  MPO: Wk 49 D1 (n=4,3,4,14) | 175.00 [87.0 to 377.0] | 180.00 [122.0 to 1340.0] | 237.00 [147.0 to 794.0] | 116.50 [43.0 to 1760.0]
  Myoglobin: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  Myoglobin: Wk 25 D1 (n=7,8,5,22) | 31.00 [19.0 to 51.0] | 31.50 [16.0 to 47.0] | 54.00 [28.0 to 112.0] | 39.50 [16.0 to 140.0]
  Myoglobin: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  Myoglobin: Wk 49 D1 (n=4,3,4,14) | 35.00 [13.0 to 47.0] | 18.00 [14.0 to 49.0] | 45.50 [31.0 to 55.0] | 45.00 [14.0 to 76.0]
  Plasmin. Activ. Inhibitor 1: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  Plasmin. Activ. Inhibitor 1: Wk 25 D1 (n=7,8,5,22) | 34.00 [13.0 to 52.0] | 45.50 [9.2 to 73.0] | 17.00 [12.0 to 41.0] | 51.50 [5.5 to 240.0]
  Plasmin. Activ. Inhibitor 1: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  Plasmin. Activ. Inhibitor 1: Wk 49 D1 (n=4,3,4,14) | 31.50 [12.0 to 42.0] | 25.00 [13.0 to 80.0] | 49.00 [14.0 to 117.0] | 52.50 [21.0 to 226.0]
  RANTES: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  RANTES: Wk 25 D1 (n=7,8,5,22) | 4.80 [1.6 to 15.0] | 5.85 [1.6 to 18.0] | 4.20 [1.8 to 13.0] | 8.80 [0.3 to 37.0]
  RANTES: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  RANTES: Wk 49 D1 (n=4,3,4,14) | 8.25 [3.4 to 14.0] | 3.20 [0.7 to 14.0] | 10.55 [0.9 to 35.0] | 6.50 [0.8 to 73.0]
  Thyroxine binding globulin Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  Thyroxine binding globulin Wk 25 D1 (n=7,8,5,22) | 38.00 [31.0 to 47.0] | 41.50 [30.0 to 75.0] | 45.00 [40.0 to 67.0] | 54.50 [33.0 to 82.0]
  Thyroxine binding globulin: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  Thyroxine binding globulin: Wk 49 D1 (n=4,3,4,14) | 42.00 [29.0 to 58.0] | 45.00 [38.0 to 51.0] | 72.50 [71.0 to 76.0] | 54.00 [37.0 to 76.0]
  TNFA: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  TNFA: Wk 25 D1 (n=7,8,5,22) | 27.00 [7.0 to 77.0] | 18.50 [7.0 to 79.0] | 25.00 [16.0 to 38.0] | 12.00 [12.0 to 319.0]
  TNFA: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  TNFA: Wk 49 D1 (n=4,3,4,14) | 32.50 [7.0 to 57.0] | 32.00 [12.0 to 51.0] | 26.50 [12.0 to 112.0] | 12.00 [12.0 to 79.0]
  TNFRT 2: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  TNFRT 2: Wk 25 D1 (n=7,8,5,22) | 33.00 [16.0 to 36.0] | 12.00 [6.2 to 53.0] | 15.00 [7.8 to 30.0] | 17.50 [5.9 to 40.0]
  TNFRT 2: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  TNFRT 2: Wk 49 D1 (n=4,3,4,14) | 28.00 [21.0 to 38.0] | 21.00 [5.5 to 29.0] | 16.00 [12.0 to 27.0] | 12.50 [3.8 to 33.0]
  VCAM1: Wk 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  VCAM1: Wk 25 D1 (n=7,8,5,22) | 2040.00 [1200.0 to 3420.0] | 1130.00 [809.0 to 2830.0] | 1690.00 [986.0 to 2770.0] | 1930.00 [984.0 to 3760.0]
  VCAM1: Wk 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  VCAM1: Wk 49 D1 (n=4,3,4,14) | 2425.00 [1200.0 to 3220.0] | 1210.00 [1160.0 to 2230.0] | 2225.00 [1410.0 to 3050.0] | 1715.00 [1030.0 to 3260.0]
  VEGF: Wk. 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  VEGF: Wk. 25 D1 (n=7,8,5,22) | 145.00 [132.0 to 429.0] | 202.50 [133.0 to 301.0] | 108.00 [64.0 to 113.0] | 168.00 [86.0 to 469.0]
  VEGF: Wks. 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  VEGF: Wks. 49 D1 (n=4,3,4,14) | 227.00 [56.0 to 286.0] | 106.00 [83.0 to 223.0] | 163.00 [87.0 to 406.0] | 217.00 [87.0 to 543.0]
  VWF: Wk. 25 D1 (n=7,8,5,22): number analyzed (Participants) | 7 | 8 | 5 | 22
  VWF: Wk. 25 D1 (n=7,8,5,22) | 135.00 [78.0 to 726.0] | 65.50 [34.0 to 140.0] | 398.00 [81.0 to 1540.0] | 156.50 [26.0 to 1230.0]
  VWF: Wk. 49 D1 (n=4,3,4,14): number analyzed (Participants) | 4 | 3 | 4 | 14
  VWF: Wk. 49 D1 (n=4,3,4,14) | 140.50 [26.0 to 385.0] | 67.00 [37.0 to 110.0] | 716.00 [25.0 to 2200.0] | 154.50 [28.0 to 2290.0]

11. Secondary Outcome: Phase Ib and Phase II: Percentage of Participants With >= 50% Reduction From Baseline in MFSAF Total Symptom Scores
Description: The 7-day modified Myelofibrosis Symptom Assessment Form (MFSAF) v2.0 is a 7-item PRO instrument based on the modified MFSAF v2.0 diary administered at specified visits. The first 6 items assess MF symptom severity at its worst as recalled in the 7 days prior to the clinic visit assessment. The symptoms measured include night sweats, itching, abdominal discomfort, pain under the ribs (left side), early satiety, & bone/muscle pain. The 7th item captures MF-related inactivity in the past 7 days prior to the clinic visit assessment. All 7 items ask subjects to record their answers on an 11-point numeric rating scale (NRS), (0 = Absent, 10 = Worst Imaginable). The first 6 items of the instrument focus on MF symptoms & are summed to create a Total Symptom score.
Time Frame: Week 24, Week 48
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDE225 400mg + INC424 10mg (Dose Escalation Phase) | LDE225 400mg + INC424 15mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 8 | 10 | 5 | 27
Percentage of participants
  Week 24 | 50.00 [15.70 to 84.30] | 40.0 [12.16 to 73.76] | 80.0 [28.36 to 99.49] | 33.3 [16.52 to 53.96]
  Week 48 | 25.00 [3.19 to 65.09] | 20.0 [2.52 to 55.61] | 80.0 [28.36 to 99.49] | 18.5 [6.30 to 38.08]

12. Secondary Outcome: Phase Ib and Phase II: Change in Total Symptom Score (TSS) From Baseline to Week 25 & Week 49 Using the MFSAF Total Symptom Scores
Description: as for outcome 11
Time Frame: Baseline, Week 25, Week 49
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- LDE225 400mg + INC424 15mg (Dose Escalation Phase): Participants who took a combination of LDE225 400mg and INC424 15mg in the dose escalation phase.
Arm/Group | LDE225 400mg + INC424 10mg (Dose Escalation Phase) | LDE225 400mg + INC424 15mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 8 | 10 | 5 | 27
scores on a scale
  Week 25 (n = 6, 7, 5, 19): number analyzed (Participants) | 6 | 7 | 5 | 19
  Week 25 (n = 6, 7, 5, 19) | -18.8 (15.20) | -14.0 (8.58) | -19.4 (6.43) | -6.5 (9.26)
  Week 49 (n = 4, 5, 4, 10): number analyzed (Participants) | 4 | 5 | 4 | 10
  Week 49 (n = 4, 5, 4, 10) | -18.5 (12.07) | -13.6 (10.43) | -21.0 (5.66) | -8.0 (14.61)

13. Secondary Outcome: Phase I and Phase II: Change in EORTC QLQ-C30 Scores From Baseline Compared to Week 24 & Week 48
Description: EORTC QLQ-C30 is the European Organization for Research & Treatment of Cancer, Quality of Life (QoL) Questionnaire & is one of the most widely used & validated instruments to measure health-related QoL in subjects with cancer. The scale includes 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning & social functioning), global health status/QoL & 9 symptom scale/items (fatigue, nausea & vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, & financial difficulties). This instrument asks the subject to respond according to the past week, with the exception of the first 5 questions that represent physical functioning & capture the subject's current status. The range of scores for all of the scales is from 0 to 100. For functional & global health status/QoL scales, higher scores indicate better QoL & level of functioning; for symptom scales, higher scores indicate greater level of symptoms or difficulties.
Time Frame: Week 24, Week 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | LDE225 400mg + INC424 10mg (Dose Escalation Phase) | LDE225 400mg + INC424 15mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 8 | 10 | 5 | 27
scores on a scale
  Glob. Health Status/Qol: Wk 25 (n=6,7,5,19): number analyzed (Participants) | 6 | 7 | 5 | 19
  Glob. Health Status/Qol: Wk 25 (n=6,7,5,19) | -2.8 (21.52) | -2.4 (21.90) | 16.7 (27.64) | 2.6 (22.75)
  Glob. Health Status/Qol: Wk 49(n=4,4,4,10): number analyzed (Participants) | 4 | 4 | 4 | 10
  Glob. Health Status/Qol: Wk 49(n=4,4,4,10) | -2.1 (23.94) | 14.6 (45.33) | -0.0 (20.41) | -3.3 (24.91)
  Phys. Func: Wk 25 (n=6,7,5,19): number analyzed (Participants) | 6 | 7 | 5 | 19
  Phys. Func: Wk 25 (n=6,7,5,19) | 15.6 (25.88) | -1.0 (14.10) | 17.3 (16.73) | 1.0 (23.74)
  Phys. Func: Wk 49 (n=4,4,4,10): number analyzed (Participants) | 4 | 4 | 4 | 10
  Phys. Func: Wk 49 (n=4,4,4,10) | 25.0 (16.67) | -10.0 (25.82) | 15.0 (22.03) | 6.0 (15.85)
  Role Func: Wk 25 (n=6,7,5,19): number analyzed (Participants) | 6 | 7 | 5 | 19
  Role Func: Wk 25 (n=6,7,5,19) | 33.3 (39.44) | -7.1 (18.90) | 16.7 (20.41) | 7.9 (32.09)
  Role Func: Wk 49 (n=4,4,4,10): number analyzed (Participants) | 4 | 4 | 4 | 10
  Role Func: Wk 49 (n=4,4,4,10) | 41.7 (21.52) | -33.3 (27.22) | 12.5 (25.00) | 10.2 (22.50)
  Emo. Func: Wk 25 (n=6,7,5,19): number analyzed (Participants) | 6 | 7 | 5 | 19
  Emo. Func: Wk 25 (n=6,7,5,19) | 25.0 (16.67) | -8.3 (31.18) | 5.6 (12.42) | 2.5 (18.61)
  Emo. Func: Wk 49 (n=4,4,4,10): number analyzed (Participants) | 4 | 4 | 4 | 10
  Emo. Func: Wk 49 (n=4,4,4,10) | 33.3 (11.79) | -12.5 (41.67) | 0.0 (15.21) | -2.5 (10.43)
  Cog. Func: Wk 25 (n=6,7,5,19: number analyzed (Participants) | 6 | 7 | 5 | 19
  Cog. Func: Wk 25 (n=6,7,5,19 | 14.6 (18.77) | -6.3 (19.80) | -3.3 (13.94) | 2.6 (18.64)
  Cog. Func: Wk 49 (n=4,4,4,10): number analyzed (Participants) | 4 | 4 | 4 | 10
  Cog. Func: Wk 49 (n=4,4,4,10) | 20.8 (15.96) | -8.3 (28.87) | 4.2 (8.33) | -5.0 (22.29)
  Soc. Func: Wk 25 (n=6,7,4,19): number analyzed (Participants) | 6 | 7 | 4 | 19
  Soc. Func: Wk 25 (n=6,7,4,19) | 8.3 (39.09) | -7.1 (18.90) | 12.5 (15.96) | -2.6 (24.38)
  Soc. Func: Wk 49 (n=3,4,4,10): number analyzed (Participants) | 3 | 4 | 4 | 10
  Soc. Func: Wk 49 (n=3,4,4,10) | 16.7 (16.67) | -4.2 (8.33) | 12.5 (25.00) | -3.3 (18.92)
  Fatigue: Wk 25 (n=6,7,5,19): number analyzed (Participants) | 6 | 7 | 5 | 19
  Fatigue: Wk 25 (n=6,7,5,19) | -20.4 (25.74) | -1.6 (26.78) | -28.9 (16.85) | -8.8 (26.86)
  Fatigue: Wk 49 (n=4,4,4,10): number analyzed (Participants) | 4 | 4 | 4 | 10
  Fatigue: Wk 49 (n=4,4,4,10) | -27.8 (6.42) | 0. (15.71) | -33.3 (18.14) | 4.4 (36.74)
  Naus & Vom: Wk 25 (n=6,7,5,19): number analyzed (Participants) | 6 | 7 | 5 | 19
  Naus & Vom: Wk 25 (n=6,7,5,19) | -5.6 (13.61) | -4.8 (18.54) | -3.3 (7.45) | -3.5 (11.89)
  Naus & Vom: Wk 49 (n=4,4,4,10): number analyzed (Participants) | 4 | 4 | 4 | 10
  Naus & Vom: Wk 49 (n=4,4,4,10) | -4.2 (15.96) | 4.2 (28.46) | 0.0 (13.61) | -10.0 (11.65)
  Pain: Wk 25 (n=6,7,5,18): number analyzed (Participants) | 6 | 7 | 5 | 18
  Pain: Wk 25 (n=6,7,5,18) | -11.1 (40.37) | -4.8 (38.14) | -26.7 (25.28) | -8.3 (21.58)
  Pain: Wk 49 (n=4,4,4,10): number analyzed (Participants) | 4 | 4 | 4 | 10
  Pain: Wk 49 (n=4,4,4,10) | 25.0 (21.52) | -8.3 (56.93) | -20.8 (25.00) | 3.3 (10.54)
  Dyspnoea: Wk 25 (n=6,7,5,19): number analyzed (Participants) | 6 | 7 | 5 | 19
  Dyspnoea: Wk 25 (n=6,7,5,19) | -33.3 (29.81) | -4.8 (29.99) | -6.7 (14.91) | -1.8 (26.00)
  Dyspnoea: Wk 49 (n=4,4,4,10): number analyzed (Participants) | 4 | 4 | 4 | 10
  Dyspnoea: Wk 49 (n=4,4,4,10) | -33.3 (27.22) | -16.7 (43.03) | 0.0 (0.00) | 6.7 (26.29)
  Insomnia: Wk 25 (n=6,7,5,19): number analyzed (Participants) | 6 | 7 | 5 | 19
  Insomnia: Wk 25 (n=6,7,5,19) | -22.2 (27.22) | 0.0 (38.49) | -33.3 (23.57) | -17.5 (34.01)
  Insomnia: Wk 49 (n=4,4,4,10): number analyzed (Participants) | 4 | 4 | 4 | 10
  Insomnia: Wk 49 (n=4,4,4,10) | -25.0 (31.91) | 8.3 (16.67) | -33.3 (27.22) | -33.3 (41.57)
  Appetite loss: Wk 25 (n=6,7,5,19): number analyzed (Participants) | 6 | 7 | 5 | 19
  Appetite loss: Wk 25 (n=6,7,5,19) | -27.8 (25.09) | 4.8 (12.60) | -13.3 (18.26) | -12.3 (29.84)
  Appetite loss: Wk 49 (n=4,4,4,10): number analyzed (Participants) | 4 | 4 | 4 | 10
  Appetite loss: Wk 49 (n=4,4,4,10) | -25.0 (41.94) | 8.3 (16.67) | -16.7 (19.25) | 0.0 (44.44)
  Constipation: Wk 25 (n=6,7,5,19): number analyzed (Participants) | 6 | 7 | 5 | 19
  Constipation: Wk 25 (n=6,7,5,19) | -11.1 (17.21) | 0.0 (0.00) | 13.3 (29.81) | 7.0 (30.59)
  Constipation: Wk 49 (n=4,4,4,10): number analyzed (Participants) | 4 | 4 | 4 | 10
  Constipation: Wk 49 (n=4,4,4,10) | -33.3 (47.14) | 0.0 (27.22) | 8.3 (16.67) | 3.3 (36.68)
  Diarrhoea: Wk 25 (n=6,7,5,19): number analyzed (Participants) | 6 | 7 | 5 | 19
  Diarrhoea: Wk 25 (n=6,7,5,19) | 5.6 (64.69) | -9.5 (16.27) | -13.3 (18.26) | -1.8 (20.71)
  Diarrhoea: Wk 49 (n=4,4,4,10): number analyzed (Participants) | 4 | 4 | 4 | 10
  Diarrhoea: Wk 49 (n=4,4,4,10) | -8.3 (16.67) | -0.0 (27.22) | 16.7 (57.74) | -3.3 (18.92)
  Fin. diff: Wk 25 (n=6,7,5,19): number analyzed (Participants) | 6 | 7 | 5 | 19
  Fin. diff: Wk 25 (n=6,7,5,19) | 16.7 (49.95) | 19.0 (32.53) | 20.0 (50.55) | 8.8 (24.45)
  Fin. diff: Wk 49 (n=4,4,4,10): number analyzed (Participants) | 4 | 4 | 4 | 10
  Fin. diff: Wk 49 (n=4,4,4,10) | 8.3 (63.10) | 25.0 (31.91) | 0.0 (27.22) | 3.3 (18.92)

14. Secondary Outcome: Phase Ib and Phase II: LDE225: PK Parameter: Racc
Description: Racc: Accumulation ratio calculated as AUC0-12h on Week 9 Day 1 divided by AUC0-12h on Week 1 Day 1 [fold]
Time Frame: 0, 0.5, 1. 1.5, 2, 4, 6, 8 hrs on Week 9 Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: ratio
Arm/Group | LDE225 400mg + INC424 10 mg (Dose Escalation Phase) | LDE225 400mg + INC424 15mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 8 | 10 | 5 | 27
ratio
  LDE225 (Week 1, Day 1) (n=0,0,0,0): number analyzed (Participants) | 0 | 0 | 0 | 0
  LDE225 (Week 9, Day 1) (n=4,6,3,13): number analyzed (Participants) | 4 | 6 | 3 | 13
  LDE225 (Week 9, Day 1) (n=4,6,3,13) | 4.60 [2.61 to 7.03] | 7.40 [4.38 to 19.6] | 10.9 [6.41 to 17.0] | 4.75 [1.84 to 20.0]

15. Secondary Outcome: Phase Ib and Phase II: INC424: PK Parameter: T1/2
Description: T1/2: Elimination half-life associated with the terminal slope (lambda_z) of a semi logarithmic concentration-time curve [time]
Time Frame: 0, 0.5, 1. 1.5, 2, 4, 6, 8 hrs on Week 1 Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: hour (h)
Arm/Group | LDE225 400mg + INC424 10 mg (Dose Escalation Phase) | LDE225 400mg + INC424 15mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 8 | 10 | 5 | 27
hour (h) | 1.81 [1.66 to 3.65] | 2.42 [1.28 to 3.14] | 2.20 [1.96 to 2.84] | 1.99 [1.34 to 3.10]

16. Secondary Outcome: Phase Ib and Phase II: INC424: PK Parameter: Vss/F
Description: Vss/F: Apparent volume of distribution at steady state after oral administration [volume]
Time Frame: 0, 0.5, 1. 1.5, 2, 4, 6, 8 hrs on Week 1 Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: Litre (L)
Arm/Group | LDE225 400mg + INC424 10 mg (Dose Escalation Phase) | LDE225 400mg + INC424 15mg (Dose Escalation Phase) | LDE225 400mg + INC424 20mg (Dose Escalation Phase) | LDED225 400mg + INC424 20mg (Dose Expansion Phase)
Number analyzed (Participants) | 8 | 10 | 5 | 27
Litre (L) | 63.7 [44.5 to 86.5] | 67.1 [41.0 to 75.7] | 53.1 [47.7 to 80.5] | 54.5 [22.9 to 102]

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 1505 days.
Groups:
- LDE225 400 mg + INC424 10 mg: Participants who took a combination of LDE225 400mg and INC424 10mg in the dose escalation phase
- LDE225 400 mg + INC424 15 mg: Participants who took a combination of LDED225 400mg and INC424 15mg in the dose escalation phase
- LDE225 400 mg + INC424 20 mg: Participants who took a combination of LDED225 400mg and INC424 20mg in the dose escalation phase
- LDE225 400 mg + INC424 20 mg (Dose Expansion): Participants who took a combination of LDED225 400mg and INC424 20mg in the dose expansion phase
- All Patients: All Patients
Arm/Group | LDE225 400 mg + INC424 10 mg | LDE225 400 mg + INC424 15 mg | LDE225 400 mg + INC424 20 mg | LDE225 400 mg + INC424 20 mg (Dose Expansion) | All Patients
All-Cause Mortality (participants affected / at risk) | 1/8 | 1/10 | 1/5 | 1/27 | 4/50
Serious Adverse Events (participants affected / at risk) | 5/8 | 6/10 | 2/5 | 13/27 | 26/50
Other Adverse Events (participants affected / at risk) | 8/8 | 10/10 | 5/5 | 27/27 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDE225 400 mg + INC424 10 mg (N=8) | LDE225 400 mg + INC424 15 mg (N=10) | LDE225 400 mg + INC424 20 mg (N=5) | LDE225 400 mg + INC424 20 mg (Dose Expansion) (N=27) | All Patients (N=50)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 2
Extramedullary haemopoiesis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 2 | 0 | 0 | 3 | 5
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0 | 3 | 5
Myoglobin blood increased (Investigations) | 0 | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDE225 400 mg + INC424 10 mg (N=8) | LDE225 400 mg + INC424 15 mg (N=10) | LDE225 400 mg + INC424 20 mg (N=5) | LDE225 400 mg + INC424 20 mg (Dose Expansion) (N=27) | All Patients (N=50)
Anaemia (Blood and lymphatic system disorders) | 5 | 4 | 4 | 16 | 29
Extramedullary haemopoiesis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2 | 3 | 7 | 15
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 0 | 4 | 9
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2
Bile acid malabsorption (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 7 | 11
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 4 | 11 | 21
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 3
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastric varices (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 8 | 12
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 3 | 2 | 1 | 5 | 11
Asthenia (General disorders) | 1 | 2 | 1 | 3 | 7
Catheter site bruise (General disorders) | 0 | 0 | 1 | 0 | 1
Early satiety (General disorders) | 0 | 1 | 0 | 1 | 2
Fatigue (General disorders) | 6 | 3 | 0 | 8 | 17
Gait disturbance (General disorders) | 0 | 0 | 0 | 2 | 2
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 1 | 0 | 1 | 3
Malaise (General disorders) | 0 | 0 | 0 | 3 | 3
Oedema peripheral (General disorders) | 2 | 2 | 0 | 1 | 5
Pyrexia (General disorders) | 0 | 2 | 2 | 7 | 11
Thirst (General disorders) | 0 | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 1 | 3
Cystitis (Infections and infestations) | 0 | 1 | 0 | 1 | 2
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 3 | 3
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 2 | 3
Influenza (Infections and infestations) | 0 | 0 | 0 | 2 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2 | 2 | 2 | 6
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 2 | 4
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 1 | 2 | 7
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 2 | 4
Urinary tract infection bacterial (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 3 | 6
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 1 | 4
Hyphaema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1 | 2 | 6
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 1 | 2 | 7
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 2 | 4
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 3 | 12 | 18
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 3 | 3
Blood prolactin increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 1 | 2
Cytomegalovirus test (Investigations) | 0 | 1 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1 | 0 | 2
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Low density lipoprotein increased (Investigations) | 0 | 0 | 2 | 1 | 3
Platelet count decreased (Investigations) | 0 | 0 | 0 | 4 | 4
Prothrombin level increased (Investigations) | 1 | 0 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 1
Weight decreased (Investigations) | 2 | 0 | 0 | 2 | 4
Weight increased (Investigations) | 1 | 1 | 0 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0 | 4 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 1 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 2
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2
Joint lock (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 6 | 4 | 18 | 31
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 2 | 8
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 9 | 13
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3 | 5
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 4 | 5
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 3 | 4 | 3 | 9 | 19
Head discomfort (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 0 | 5 | 8
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 2 | 3
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 1 | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0 | 1 | 2
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2 | 2
Depression (Psychiatric disorders) | 0 | 2 | 0 | 1 | 3
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 2 | 4
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 5 | 11
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 3 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 7 | 3 | 12 | 25
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 3 | 5
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 4
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 4
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 1 | 0 | 1 | 3
Hypertension (Vascular disorders) | 0 | 1 | 1 | 5 | 7
Intermittent claudication (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 1 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Please refer to detailed description regarding reason for early termination of study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie. data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-08-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT01787552/SAP_000.pdf
  • Study Protocol (2015-02-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT01787552/Prot_001.pdf